CLINICAL TRIAL: NCT03341234
Title: Analgesic Efficiency of Superficial Serratus Plane Block for Modified Radical Mastectomy and Axillary Lymph Node Disection: Randomized Controlled Study
Brief Title: Superficial Serratus Plane Block for Modified Radical Mastectomy and Axillary Lymph Node Disection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Superficial SPB
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Analgesia; Pain, Postoperative; Opioid Consumption
Keywords: Superficial Serratus Plane Block; Modified Radical Mastectomy; Axillary Lymph Node Disection; bupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Sodium Chloride; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group SPB (Active Comparator): Ultrasound guided serratus plane block with 30 ml %0,25 bupivacaine
  Interventions: Drug: Bupivacaine; Device: Ultrasound
- Group Control (Active Comparator): Ultrasound guided sham block with 2 ml saline subcutaneously
  Interventions: Drug: Saline; Device: Ultrasound

INTERVENTIONS:
Drug: Bupivacaine — 30 ml %0,25 bupivacaine
  Arms: Group SPB
Drug: Saline — 2 ml saline subcutaneously
  Arms: Group Control
Device: Ultrasound — Ultrasound guided block

SUMMARY:
Breast cancer is the most common type of cancer in women. Mastectomy and axillary lymph node disection are commonly performed as part of the cancer management. This surgery can cause significant postoperative pain. The serratus plane block (SPB) has been described for analgesia of the hemithorax and reported for many cases such as thoracoscopy, shoulder arthroscopy, breast surgery and axillary lymph node dissections. Serratus plane block may be a viable alternative to current regional anaesthetic techniques such as thoracic paravertebral and central neuraxial blockade.

The aim of this study is to determine effectiveness of ultrasound guided superficial serratus plane block in patients undergoing modified radical mastectomy and axillary lymph node dissection surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients undergoing Modified Radical Mastectomy and Axillary Lymph Node Disection

Exclusion Criteria:

* chronic pain, bleeding disorders, renal or hepatic insufficiency,patients on chronic non-steroidal anti-inflammatory medications

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | First 24 hours total opioid consumption
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | postoperative first hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at first hour postoperatively.
Visual analog pain score | postoperative second hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at second hour postoperatively.
Visual analog pain score | postoperative 4th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 4th hour postoperatively.
Visual analog pain score | postoperative 8th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 8th hour postoperatively.
Visual analog pain score | postoperative 12th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 12th hour postoperatively.
Visual analog pain score | postoperative 24th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 24th hour postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Training and Research Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Ahiskalioglu A, Alici HA, Yayik AM, Celik M, Oral Ahiskalioglu E. Ultrasound guided serratus plane block for management of acute thoracic herpes zoster. Anaesth Crit Care Pain Med. 2017 Oct;36(5):323-324. doi: 10.1016/j.accpm.2017.01.008. Epub 2017 Mar 21. No abstract available. PMID 28336228